CLINICAL TRIAL: NCT00005086
Title: A Phase II Trial of "Sequential Doublets" Chemotherapy in Patients With Locally Advanced or Metastatic Bladder Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Stage IV Locally Advanced or Metastatic Bladder Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11203; UCCRC-11203; NCI-G00-1733
Record Dates: First submitted 2000-04-06; First posted 2003-05-16 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Bladder Cancer
Keywords: stage IV bladder cancer; transitional cell carcinoma of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Docetaxel; Gemcitabine; Methotrexate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): Methotrexate will be given as a short infusion (introduced into a vein) for approximately 5 minutes on the first day (day 1). ). A week later (day 8), both methotrexate and docetaxel will be given the same way, but this will take about 1 hour. The first course of treatment consists of receiving treatment on day 1 and day 8 every 21 days for 9 weeks. X-rays or scans will then be performed to determine if your tumor is shrinking. You will then start treatment with gemcitabine and cisplatin. On the first day (day 1), you will receive both cisplatin and gemcitabine into your vein. A week later (day 8), you will receive only gemcitabine as an infusion into your vein over 100 minutes and no additional intravenous fluid will be required on that day. This second course of treatment consists of receiving treatment on day 1 and day 8 every 21 days for 9 weeks.
  Interventions: Drug: cisplatin; Drug: docetaxel; Drug: gemcitabine hydrochloride; Drug: methotrexate

INTERVENTIONS:
Drug: cisplatin
Drug: docetaxel
Drug: gemcitabine hydrochloride
Drug: methotrexate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy in treating patients who have stage IV locally advanced or metastatic bladder cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate to the combination of docetaxel and methotrexate followed by gemcitabine and cisplatin in patients with stage IV locally advanced or metastatic, previously untreated, transitional cell carcinoma of the urothelium.
* Assess the toxicities of this sequential regimen in this patient population.
* Assess time to event efficacy measures including time to disease progression, duration of response, and overall survival in these patients treated with this sequential regimen.

OUTLINE: Patients receive methotrexate IV on days 1 and 8 and docetaxel IV over 1 hour on day 8 every 3 weeks for 9 weeks. Patients then receive cisplatin IV over 2 hours on day 1 and gemcitabine IV over 100 minutes on days 1 and 8 every 3 weeks for 9 weeks. This 18 week sequential regimen constitutes 1 full course. Treatment continues in the absence of unacceptable toxicity or disease progression.

Patients are followed until death or until 2 years after study entry, whichever comes first.

PROJECTED ACCRUAL: A total of 18-46 patients will be accrued for this study within 9-24 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV locally advanced or metastatic transitional cell carcinoma of the urothelium that is not amenable to curative surgery or radiotherapy

  * T4b or N2 or N3 or M1
  * No pure adenocarcinomas, pure squamous carcinomas, or small cell carcinoma
* Evaluable or bidimensionally measurable disease If only single lesion, must not be within portal of prior irradiation
* No active CNS metastases

  * Adequately treated CNS metastases eligible provided stable for 8 weeks following therapy and no longer requires steroids or antiseizure medication
* No clinically significant pleural effusions or ascites unless drained prior to administration of methotrexate

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* CALGB 0-1

Life expectancy:

* At least 12 weeks

Hematopoietic:

* Granulocyte count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 9.0 g/dL (transfusion allowed)

Hepatic:

* Bilirubin less than 1.5 mg/dL
* SGOT less than 2.5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 50 mL/min

Cardiovascular:

* No uncontrolled cardiac disease (e.g., congestive heart failure, arrhythmia, or angina)

Pulmonary:

* No uncontrolled pulmonary disease (e.g., chronic obstructive pulmonary disease)

Other:

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after study participation
* No concurrent active infection
* No known hypersensitivity to docetaxel, methotrexate, cisplatin, gemcitabine, filgrastim (G-CSF), oprevelkin, or any component of these products
* No serious concurrent medical disorder
* No medical or psychiatric conditions that would compromise consent or preclude completion of study
* No other malignancy within the past 3 years except:
* Carcinoma in situ of the cervix
* Adequately treated nonmelanoma skin cancer
* Stage I or II prostate cancer provided adequate local therapy (surgery or radiation) has been administered and PSA is less than 1.0 ng/mL
* No preexisting peripheral neuropathy grade 2 or greater

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior systemic chemotherapy for metastatic disease
* At least 6 months since prior neoadjuvant or adjuvant chemotherapy
* No other concurrent chemotherapy

Endocrine therapy:

* No concurrent steroids

Radiotherapy:

* See Disease Characteristics
* No concurrent radiotherapy

Surgery:

* See Disease Characteristics
* At least 3 weeks since prior major surgery and recovered

Other:

* No other concurrent investigational drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 1999-08; Primary Completion 2002-08 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Safety and toxic effects of giving docetaxel and methotrexate followed by gemcitabine and cisplatin | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (4):
- United States (4):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana